CLINICAL TRIAL: NCT00459550
Title: A Randomised, Single-Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, Immunogenicity, Pharmacokinetics and Pharmacodynamics of Intravenous Infusion of GSK933776 in Patients With Alzheimer's Disease.
Brief Title: A Clinical Study to Assess Single and Repeat Doses of a New Medication (GSK933776) in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 106006
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; First Time in Human (FTIH) Study
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Experimental): Part A will be a single-blind, single dose, placebo controlled, dose escalation study in up to five consecutive cohorts of Alzheimers Disease subjects. Each subject will receive a single infusion of GSK933776 or placebo. The dose for the first cohort will be 0.001 mg/kg. The proposed nominal doses for subsequent cohorts are 0.01, 0.1, 0.5 and 3 mg/kg, but these may be altered based on the outcome of the safety, tolerability, pharmacodynamic and pharmacokinetic data of the preceding group(s). The maximum possible dose will be 20 mg/kg, although the planned top dose is 18 mg/kg
  Interventions: Drug: GSK933776; Drug: Placebo to match GSK933776
- Part B (Experimental): Part B will be a single-blind, repeat dose, placebo controlled dose escalation design. It is proposed that there will be initially 3 cohorts of AD subjects. However up to 5 cohorts may be recruited if required in order to characterise GSK933776 fully.Each cohort will consist of eight subjects (six active, two placebo) who will each receive a maximum of three infusions of GSK933776 or placebo. Dosing in Part B may proceed in parallel with Part A following satisfactory review of minimum data sets as below:
  First cohort in Part B: at least 3 weeks' data from the Part A dose that is the same dose level as that planned for Part B Second cohort in Part B: at least 3 weeks PK data and 8 weeks safety data following the first dose from all the subjects on active treatment in the preceding Part B cohort plus a satisfactory outcome of the PIB Subsequent cohorts in Part B: at least 3 weeks PK data and 8 weeks safety data follow
  Interventions: Drug: GSK933776; Drug: Placebo to match GSK933776

INTERVENTIONS:
Drug: GSK933776 — Part A planned doses cohort 1 to cohort 3 0.001 mg/kg, 0.01 mg/kg and 0.1 mg/kg.
  Part B planned doses cohort 4 to cohort 7 0.1 mg/kg, 1mg/kg, 3mg/kg and 10 mg/kg
  Other Names: GSK933776A
Drug: Placebo to match GSK933776 — Part A first 2 cohorts 5 patients per cohort 2 placebo and 3 active third cohort part A 2 placebo 6 active. Part B 8 patients per cohort 2 placebo 6 active.

SUMMARY:
A study to investigate the safety and tolerability of both single and multiple intravenous administration of GSK933776 in patients with Alzheimer's Disease.

ELIGIBILITY:
Inclusion criteria:

* Male or female subject with a clinical diagnosis of probable Alzheimer's disease
* Subject has mild AD with Mini Mental State Examination (MMSE) score 18-26 inclusive at the screening visit.
* Age between 55 and 80 years.
* Female subjects must be post-menopausal or surgically sterile.
* Male subjects whose partner is of child-bearing potential or have been menopausal for <2 years must use an adequate form of contraception.
* Subject has the ability to comply with procedures for cognitive and other testing & is fluent in the language used for the administration of the cognitive tests.
* Subject lives with (or has substantial periods of contact with) a permanent caregiver who is willing to oversee the subject's compliance with protocol-specified procedures and study medication, and report on subject's status.
* Subject has provided full written informed consent prior to the performance of any protocol-specified procedure.
* Caregiver has provided a full written informed consent on his/her own behalf prior to the performance of any protocol-specified procedure.

Exclusion criteria:

* History and/or evidence of any other central nervous system (CNS) disorder that could be interpreted as a cause of dementia.
* Subjects currently living in a nursing home.
* Subjects who are unable to provide informed consent due to cognitive status
* Screening brain MRI with 1 or more of the following conditions: not consistent with AD, evidence of other CNS conditions, shows more than minimal vascular changes, more than 3 microhaemorrhage lesions.
* Focal findings on the neurological exam.
* Any contraindication to lumbar puncture.
* History or evidence of significant psychiatric illness such as schizophrenia or bipolar affective disorder or significant neurological disease other than AD.
* TIA/stroke in the last 3 years, type 1 or type 2 diabetes mellitus, active cardiovascular disease, or other uncontrolled risk factors for stroke.
* Current or recent drug or alcohol abuse or dependence or recent or remote history of the same if that could be a contributing factor to the dementia.
* History or evidence of any significant autoimmune disease or disorder.
* History of seizures (excluding febrile seizures in childhood), current blood clotting or bleeding disorder or conditions that predispose to these (e.g. cancer), current clinically significant systemic illness or significant infection within 30 days that is likely to result in deterioration of the subject's condition or affect the subject's safety during the study.
* History of cerebral amyloid antiopathy and/or hypertensive cerebral haemorrhage or with a known risk of intercerebral haemorrhage/microhaemorrhage.
* Treatment which cholinesterase inhibitors, memantine or selegiline unless the therapy was instituted at least 3 months prior to the administration of GSK933776, at a stable dosage in the 2 months prior and the same regimen will be continued for the duration of the trial and the subject is free from any clinically significant side effects attributable to the drug.
* Subjects who have discontinued cholinesterase inhibitors, memantine, cognitive enhancing agents, or drugs that potentially affect cognition in the 60 days prior to screening.
* Unless maintained on a stable dose regimen for at least 30 days prior to screening, any other medications with the potential to affect cognition.
* Use of drugs with platelet anti-aggregant or anti-coagulant properties (excluding the use of aspirin 325 mg/day or less), anticonvulsants for seizures or narcotic medication.
* History of or current chronic use of systemic steroids or other immunosuppressants.
* Prior participation in clinical investigations involving therapeutic monoclonal antibodies or proteins derived from monoclonal antibodies or any investigations of treatments or use of experimental medications for AD or any other investigational medication or device within 60 days prior to screening or within 5 half-lives of use of such a medication prior to screening, whichever is longer.
* Contraindications for MRI: pacemaker, aneurysm clips, artificial heart valves, other metal foreign body, claustrophobia, etc.
* Smoking more than 20 cigarettes or equivalent per day.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03-12 (Actual); Primary Completion 2011-05-30 (Actual); Study Completion 2011-05-30 (Actual)

PRIMARY OUTCOMES:
Adverse events. Changes suggesting potential adverse events detected in the physical & neurological examination, brain MRI, cognitive status, laboratory parameters, ECG & vital signs. | 12 weeks for Part A; 34 weeks in Part B

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters of GSK933776. Pharmacodynamic effects of GSK 933776. CSF detectable levels of GSK933776. Effects of GSK933776 on plasma and CSF biomarkers. Titre & neutralising activity of anti-GSK933776 antibodies. Exploratory PET scan | 12 weeks for Part A; 34 weeks in Part B

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Australia (3):
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Heidelberg Heights, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
- GSK Investigational Site, Lørenskog, Norway
- Sweden (3):
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Mölndal
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Andreasen N, Simeoni M, Ostlund H, Lisjo PI, Fladby T, Loercher AE, Byrne GJ, Murray F, Scott-Stevens PT, Wallin A, Zhang YY, Bronge LH, Zetterberg H, Nordberg AK, Yeo AJ, Khan SA, Hilpert J, Mistry PC. First administration of the Fc-attenuated anti-beta amyloid antibody GSK933776 to patients with mild Alzheimer's disease: a randomized, placebo-controlled study. PLoS One. 2015 Mar 19;10(3):e0098153. doi: 10.1371/journal.pone.0098153. eCollection 2015. PMID 25789616
- See also: Results for study 106006 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/106006?search=study&study_ids=106006#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 106006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register